CLINICAL TRIAL: NCT01808820
Title: Dendritic Cell Vaccine For Malignant Glioma and Glioblastoma Multiforme in Adult and Pediatric Subjects
Brief Title: Dendritic Cell (DC) Vaccine for Malignant Glioma and Glioblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Macarena De La Fuente, MD (Other)
Responsible Party: Sponsor-Investigator, Macarena De La Fuente, MD, Assistant Professor of Clinical, University of Miami
Organization: University of Miami (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20120750
Record Dates: First submitted 2013-03-06; First posted 2013-03-11 (Estimated); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Malignant Glioma; Glioblastoma Multiforme; Anaplastic Astrocytoma; High Grade Glioma
Keywords: HGG; Dendritic Cell Vaccine; DC Vaccine; Leukapheresis
MeSH Terms: conditions — Glioma; Glioblastoma; Astrocytoma | interventions — lentiviral minigene vaccine of COVID-19 coronavirus; Imiquimod; Leukapheresis; Blood Component Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Safety Pilot: DC Vaccine/Lysate (Experimental): Participants in this group will undergo leukapheresis after standard of care surgical tumor resection. Leukapheresis will be used to obtain peripheral blood mononuclear cells (PBMC) from which the dendritic cells (DC) will be obtained. Retrieved DC will be used as a vaccine once weekly on Weeks 1-4 within 3 weeks from end of leukapheresis. Participants will also receive Imiquimod, which will be applied one evening prior to DC dose for 8 hours then for 8 hours each of the next two evenings. Enrollment of participants in the Pilot group will be staggered until the second participant has no treatment limiting toxicities. For the first five subjects to be enrolled in the pilot, the administration of DC to each subject will be delayed until the prior subject has received the second administration of DC. Participants will also receive Lysate of tumor administered every 4 weeks + 3 days on Weeks 8, 12, 16 and 28 (+ / - 3 days).
  Interventions: Biological: Dendritic Cell Vaccine; Biological: Tumor Lysate; Drug: Imiquimod; Procedure: Leukapheresis
- Expansion Cohort: DC Vaccine/Lysate (Experimental): Participants in this group will undergo leukapheresis within after standard of care surgical tumor resection. Leukapheresis will be used to obtain peripheral blood mononuclear cells (PBMC) from which the dendritic cells (DC) will be obtained. Retrieved DC will be used as a vaccine once weekly on Weeks 1-4 within 3 weeks from end of pheresis. Participants will also receive Imiquimod, which will be applied one evening prior to DC dose for 8 hours then for 8 hours each of the next two evenings. Participants will also receive Lysate of tumor administered every 4 weeks + 3 days on Weeks 8, 12, 16 and 28 (+ / - 3 days).
  Interventions: Biological: Dendritic Cell Vaccine; Biological: Tumor Lysate; Drug: Imiquimod; Procedure: Leukapheresis

INTERVENTIONS:
Biological: Dendritic Cell Vaccine — Between 1.2 to 12 million DC per dose administered once a week via intradermal injection for 4 weeks.
  Other Names: DC Vaccine
Biological: Tumor Lysate — Post-DC Vaccine therapy. Up to 1.5 mg of Lysate of tumor per dose administered via intradermal injection at intervals defined by study protocol.
  Other Names: Lysate of Tumor; Lysate Boost
Drug: Imiquimod — 5% topical cream applied to vaccine site before and after administrations of DC vaccine or lysate
  Other Names: Aldara
Procedure: Leukapheresis — Baseline, post-surgery blood draw via catheter to obtain peripheral blood mononuclear cells (PBMCs) from which Dendritic cells will be obtained.
  Other Names: Pheresis

SUMMARY:
The purpose of this research study is to evaluate an investigational vaccine using patent-derived dendritic cells (DC) to treat malignant glioma or glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 13 years and ≤ 99 years.
2. (2a) Relapse of high grade glioma (anaplastic astrocytoma World Health Organization (WHO) grade III or glioblastoma multiforme WHO grade IV), histologically proven at first stage of disease (radiological evidence for recurrence suffices); OR (2b) Relapse of glioma, which was grade II at initial diagnosis, but which is grade III or IV at relapse based on radiological or pathological criteria.
3. Total or subtotal resection of tumor mass, confirmed by assessment by the neurosurgeon and by postoperative MRI scan within 72 hours after surgery. The post-operative assessment should demonstrate residual tumor less than or equal to 2 cm^3 as judged by surgeon and on MRI the tumor should only show linear contrast enhancement at the border of the resection cavity or nodule less than 2 cm^3.
4. No radiotherapy and/or chemotherapy received for at least 1 month before first DC vaccination is to be administered
5. No treatment with corticosteroids or salicylates for at least 1 week before first vaccination. Corticosteroid therapy should be rapidly weaned within 1-2 weeks after surgery.
6. Life expectancy > 3 months.
7. Written consent by patient or parent(s) (if patient is < 18 years) on an institutional review board (IRB)-approved informed consent form prior to any study-specific evaluation. Assent is required from children as per University of Miami (UM) IRB guidelines. Subject must be capable of understanding the investigational nature, potential risks and benefits of the study and able to provide valid informed consent.
8. Adequate organ function (to be measured at enrollment)

   * Absolute neutrophil count (ANC) ≥ 0.75 10*3/µl
   * Lymphocytes ≥ 0.5 10*3/µl
   * Platelets ≥ 75 10*3/µl
   * Hemoglobin ≥ 9 g/dL
   * Aspartate transaminase (AST)/Alanine transaminase (ALT) ≤ 2.5 X upper limit of normal (ULN); if liver metastases, ≤ 5 X ULN
   * Serum Creatinine ≤ 1.5 X ULN
   * Total Bilirubin ≤ 3 X ULN
   * Albumin > 2 g/dL
9. Subjects must agree to use adequate method of contraception or abstinence throughout and up to 4 weeks after the study treatment completion.
10. Karnofsky score 70 or higher or Eastern Cooperative Oncology Group (ECOG) status of 0 or 1.

Exclusion Criteria:

1. Pregnancy.
2. Breast feeding females.
3. Any concomitant participation in other therapeutic trials.
4. Virus serology positive for HIV (testing is not required in the absence of clinical suspicion).
5. Documented immunodeficiency or autoimmune disease.
6. Mandatory treatment with corticosteroids or salicylates in the week prior to first vaccination.
7. Other active malignancies.
8. Patients with unresectable tumors, for instance pontine gliomas, are excluded.
9. Refusal to use adequate contraception for fertile patients (females and males) during the study and for 30 days after the last dose of study treatment.
10. Any serious or uncontrolled medical or psychiatric condition that in the opinion of the investigator makes the patient not able to participate in the study.
11. Application of gliadel wafers within the prior 4 months or a plan to place gliadel wafers at the time of resection for tumor acquisition for study.

Ages: 13 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-08-21 (Actual); Primary Completion 2018-11-07 (Actual); Study Completion 2022-07-16 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events | Up to Week 32 (30 days after last dose of protocol therapy)
  Adverse Events will be evaluated using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 4.0 by treating physician

SECONDARY OUTCOMES:
Rate of Overall Survival (OS) in Study Participants | Up to Week 80 (5 years post therapy)
  Rate of overall survival in study participants receiving protocol therapy. Overall survival is defined as the time elapsed from the start of treatment until death. For surviving patients, follow-up will be censored at the date of last contact.
Rate of Progression-Free Survival (PFS) in Study Participants | Up to Week 80 (5 years post therapy)
  Rate of prolonged progression-free survival in study participants receiving protocol therapy. Progression-Free Survival (PFS) is defined as the time elapsed from the start of treatment to the date of documented progression or death, whichever comes first. For surviving patients without progression who begin alternative treatment, PFS will be censored at the last date of documented progression-free status prior to starting alternative treatment. Similarly, losses to follow up will be censored at the last date of documented progression-free status.
Change in MDSC Levels | Baseline, Up to Week 28
  Immune response will be reported as the change in Myeloid Derived Suppressor Cell (MDSC) levels from blood samples
Change in blood counts | Baseline, Up to Week 28
  Measurement of immune response will be reported as the change in red and white blood counts from blood samples evaluated in million cells/microliter
Comparison of clinical parameters associated with outcomes in study participants to patients on other DC/Imiquimod studies. | Up to 5 years Post-Therapy
  To demonstrate if the clinical parameters associated with outcomes described for patients on other DC / imiquimod protocols hold for subjects treated on this study.
Proportion of participants completing intervention. | Up to Week 28
  Proportion of participants able to receive all administrations of DC vaccine and those who are able to receive all administration of DC vaccine and lysate will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Macarena De La Fuente, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No